CLINICAL TRIAL: NCT01694355
Title: The Impact of Severe Vitamin D Deficiency and Its Correction on Bone Mineral Density (BMD) in Postmenopausal Women
Acronym: Vitamin D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Merav Fraenkel, Senior Endocrinologist, Soroka University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sor0089-12-ctil; SCRC12008 (Other: Soroka Clinical Research Center (SCRC))
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D treatment (Experimental): We assume that among postmenopausal women, Vitamin D treatment will improve bone mineralization and will cause a rapid increase in BMD.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D

SUMMARY:
It is well known that postmenopausal women are at risk for osteoporosis. The study hypothesis is that vitamin D deficiency (≤17.5nmol/L) is frequently associated with osteomalacia and will cause low BMD estimation in DXA scan due to insufficient bone mineralization.

We assume that among these postmenopausal women, Vitamin D treatment will improve bone mineralization and will cause a rapid increase in BMD. According to the results, bisphosphonates therapy may be an unnecessary treatment.

The objective of this study is to evaluate the impact of severe vitamin D deficiency and its correction on Bone Mineral Density (BMD) in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent.
2. Female age 55-70
3. At least 2 years past menopause
4. 25(OH)D≤ 17.5nmol/L (≤7 ng/ml)

Exclusion Criteria:

1. Vitamin D levels > 30nmol/L in the past 2 years 2. Creatinine > 1.2%mg 3. Calcium ≥ 10.2mg/dl 4. Current or previous vitamin D treatment over 2 weeks 5. Previous vitamin D treatment over 2 months in the past 2 years 6. BMI>35 or BMI<20 7. Menopause before age 45 8. Type 1 diabetes 9. Concomitant disease:

1. Mal-absorptive diseases (Cystic Fibrosis, Crohn's, gastric bypass surgery, celiac disease)
2. Rheumatoid arthritis
3. Nephrotic syndrome
4. Chronic renal failure
5. Primary hyperparathyroidism
6. Hyperthyroidism
7. Malignancies excluding skin cancers (within the last 5 years)
8. Kidney stones or history of renal colic 10. Medications:
9. Steroids use (past or present)
10. Anti rejection drugs in the last 5 years
11. Anticonvulsant (carbamezapine, hydantoin, Phenobarbital etc) in the last 5 years
12. Any anti osteoporotic medication: Prolia, Bisphosphonates, Teriperatide, Evista, Protelos, (past or present)
13. Post menopausal HRT (in the last 10 years)
14. Aromatase inhibitors: Femara, Arimadex (past or present)
15. Current use of PPIs (lanton, controloc, zoton, omepradex etc)
16. Current or past use of anti depressant SSRI (favoxil,cipralex etc)

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in BMD (Z score) following 10 months of vitamin D supplementation | 10-14 months
  Will be measured at 3 time points (repeated measures):at baseline visit, after 3-4 months and after 10 months of treatment

SECONDARY OUTCOMES:
To examine the effect of increasing vitamin D levels on other objective parameters such as PTH, calcium, phosphorus and other subjective parameters such as muscle weakness, according to comparison between baseline visit and end of study visit. | 10-14 months
  Will be measured at 3 time points (repeated measures):at baseline visit, after 3-4 months and after 10 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No